CLINICAL TRIAL: NCT00815724
Title: Distributed Asthma Learning Initiative
Brief Title: Evaluating a Distance Learning Asthma Education Program for Pediatricians (The DALI Study)
Acronym: DALI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 621; R01HL070771 (NIH)
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Asthma
Keywords: Daily Inhaled Corticosteroids; Distributed Learning; E-learning
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will take part in a distance learning group.
  Interventions: Behavioral: Distributed Asthma Learning Initiative (DALI) distance learning program
- 2 (No Intervention): Participants in the control group will not receive any study materials or take part in any study activities.

INTERVENTIONS:
Behavioral: Distributed Asthma Learning Initiative (DALI) distance learning program — Participants will take part in two Webinar teleconferences, have access to an interactive Web site, and receive a CD-ROM of study materials and a toolkit.
  Arms: 1

SUMMARY:
The National Heart, Lung, and Blood Institute (NHLBI) has established guidelines for treating people with asthma. This study will evaluate the effectiveness of a distance learning program that aims to educate doctors on these guidelines, specifically the use of inhaled corticosteroids to treat asthma in pediatric patients.

DETAILED DESCRIPTION:
Asthma is a long-term lung disease that affects more than 22 million people in the United States. Symptoms include wheezing, chest tightness, shortness of breath, and coughing. Inhaled corticosteroids are a common medication used to treat asthma. NHLBI has established guidelines for doctors to reference when treating people with asthma. Study researchers previously evaluated a distance learning program aimed to educate doctors on the NHLBI guidelines and to improve pediatrician adherence to the guideline recommendations for the use of daily inhaled corticosteroids for persistent asthma in pediatric patients. This pilot study will evaluate a new version of the distance learning program. By using a distance learning program rather than a traditional face-to-face educational program, participants will be able to complete the program on their own schedule, and this flexibility may result in increased interest in the program. The purpose of this study is to evaluate the effectiveness of the new distance learning program on changing pediatricians' behavior, attitudes, and knowledge regarding the NHLBI guidelines for the use of inhaled corticosteroids to treat pediatric patients with asthma.

This study will enroll pediatricians. Participants will be randomly assigned to either the distance learning group or a control group. At baseline, all participants will complete questionnaires. Participants in the control group will not take part in any of the educational activities. Participants in the distance learning group will take part in a 1-hour Webinar, or teleconference, that will provide an orientation to the program and discuss the importance of the NHLBI guidelines. At any time between the first Webinar and a 6-week follow-up Webinar, participants will log into the study Web site and complete a training module that aims to educate participants on common barriers to prescribing daily inhaled corticosteroids. As an alternative to the Web site, participants may choose to view the training module on a CD-ROM. Six weeks after the first Webinar, participants will take part in a follow-up Webinar. At this time, study researchers will answer participants' questions and provide a program review. The Web site and study materials will remain available to participants in the distance learning group for 6 months after the follow-up Webinar; a list serve will also be made available to participants. At 1 and 6 months after the follow-up Webinar, all participants will complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Board-eligible pediatricians involved in direct primary care for children
* Has access to a Windows or Macintosh computer with either a CD-ROM drive or Internet access
* Has access to a telephone for teleconference calls
* Willing to take part in the DALI educational seminar if assigned to the intervention group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change in physician asthma knowledge, attitudes, and treatment behavior | Measured at Months 1 and 6
Learner satisfaction | Measured at Months 1 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Cabana, MD, MPH, Principal Investigator — University of California, San Francisco; Tao Le, MD, Principal Investigator — University of Louisville
Locations (1):
- University of California, San Francisco, San Francisco, California, United States